CLINICAL TRIAL: NCT07110441
Title: A Phase 1, Open Label Study to Assess Pharmacokinetics, Safety and Tolerability of G1090N in Healthy Subjects
Brief Title: Pharmacokinetic Study on G1090N (Nitazoxanide) Capsules in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: G1090N_P1_25_1
Record Dates: First submitted 2025-07-25; First posted 2025-08-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-09

CONDITIONS: Acute-on-Chronic Liver Failure
Keywords: Acute-on-Chronic Liver Failure; ACLF; G1090N, Tizoxanide, Nitazoxanide, Pharmacokinetics, Healthy volunteer
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- G1090N 300 mg (Experimental): Subjects will recieve a single dose of G1090N
  Interventions: Drug: Single Dose G1090N
- G1090N 600 mg (Experimental): Subjects will recieve single and multiple doses of G1090N
  Interventions: Drug: Single Dose G1090N; Drug: Multiple dosing of G1090N
- G1090N 900 mg (Experimental): Subjects will recieve single and multiple doses of G1090N
  Interventions: Drug: Single Dose G1090N; Drug: Multiple dosing of G1090N
- G1090N 1200 mg (Experimental): Subjects will recieve single and multiple doses of G1090N
  Interventions: Drug: Single Dose G1090N; Drug: Multiple dosing of G1090N

INTERVENTIONS:
Drug: Single Dose G1090N — Subjects will receive single ascending doses of G1090N up to 1200mg.
Drug: Multiple dosing of G1090N — Subjects will receive multiple ascending doses of G1090N up to 1200mg twice daily for 7 consecutive days.
  Arms: G1090N 1200 mg; G1090N 600 mg; G1090N 900 mg

SUMMARY:
A Phase 1, Open-Label Study to Assess Pharmacokinetics, Safety and Tolerability of G1090N in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy subjects with absence of clinically relevant abnormalities as determined by the Investigator or medically qualified designee based on a detailed medical history and complete physical examination;
* 2. Clinical laboratory test results for liver and renal function within the normal reference range. For all other clinical laboratory parameters, results outside the normal reference range to be confirmed by the Investigator and the Sponsor as not clinically significant;
* 3. Male or female subjects ≥18 and ≤55 years of age with a minimum body weight of 50 kg and a body mass index of ≥18.0 to ≤30.0 kg/m2 at the time of signing the informed consent form (ICF);
* 4. Subjects willing and able to comprehend and sign informed consent and to comply with the requirements of this study.

Exclusion Criteria:

* 1. Significant history or clinical manifestation of any metabolic (including thyroid), allergic, dermatological, hepatic (including Gilbert's syndrome), renal, hematological, pulmonary, cardiovascular (including any prior history of cardiomyopathy or cardiac failure), gastrointestinal, neurological, or psychiatric disorder;
* 2. Experienced an acute illness within 14 days of SCR;
* 3. Positive serologic test for hepatitis B surface antigen, or for hepatitis C virus antibody, or human immunodeficiency virus I and II at SCR; positive coronavirus disease 2019 test at Day -1 of Part 1 or Part 2;
* 4. Frequent headaches (more than twice a month) and/or migraines, recurrent nausea and/or vomiting, or diarrhea;
* 5. Smokers, defined as having used tobacco- or nicotine-containing products within 6 months prior to SCR;
* 6. Out-of-range vital signs at rest (ie, supine for at least 5 minutes) at SCR and Day -1 of Part 1 and Part 2, defined as:

  1. Systolic blood pressure (SBP) <90 mm Hg or >140 mm Hg;
  2. Diastolic blood pressure (DBP) <50 mm Hg or >90 mm Hg;
  3. Pulse rate <50 bpm or >90 bpm; For these parameters, out-of-range values that are not clinically significant (as determined by the Investigator) may be repeated twice during SCR and the subject may be enrolled if at least one repeated value is within the range noted above;
* 7. Symptomatic hypotension at SCR, regardless of the decrease of blood pressure, or asymptomatic postural hypotension defined by a decrease in SBP ≥20 mm Hg or DBP ≥10 mm Hg within 3 minutes when changing from the supine to the standing position;
* 8. Out-of-range 12-lead electrocardiogram (ECG) recordings at SCR defined as:

  1. PR ≤120 ms or ≥220 ms;
  2. QRS >120 ms;
  3. QT interval corrected for heart rate using Fridericia's method ≥450 ms; For these parameters, out-of-range values that are not clinically significant (as determined by the Investigator) may be repeated twice during SCR and Day -1 and the subject may be enrolled if at least 1 repeated value is within the normal ranges noted above; Subjects must also have no sign of any clinically significant irregularity in heart rhythm.
* 9. Use of any prescription or nonprescription drugs or substances (including vitamins and dietary or herbal supplements) within 30 days or 5 half-lives, if known, of the respective drug or substance, whichever is longer, prior to investigational medicinal product (IMP) administration, unless deemed acceptable by the Investigator and Sponsor;
* 10. Vaccination with a live vaccine within 6 months prior to first dosing or vaccination with an inactivated vaccine (eg, inactivated influenza vaccines or severe acute respiratory syndrome coronavirus 2 vaccines) within 30 days prior to first dosing;
* 11. Receipt of NTZ, or any investigational product within 30 days, or 5 half-lives, if known, of the respective investigational product, whichever is longer, prior to SCR;
* 12. History of alcohol consumption defined as >30 g pure alcohol/day for men, and >20 g pure alcohol/day for women within the last year, or any alcohol consumption within 48 hours prior to SCR or Day -1 for Part 1 and Part 2;
* 13. Consumption of caffeine- or xanthine-containing products (>4 cups or glasses per day of eg, coffee, tea, cola drinks, and chocolate) within 48 hours prior to SCR or Day -1 for Part 1 and Part 2;
* 14. Subjects following a vegan or vegetarian diet or any other dietary restrictions;
* 15. Strenuous exercise within 24 hours prior to SCR or Day -1 for Part 1 and Part 2;
* 16. Blood donation or blood loss (excluding volume drawn at SCR) of 50 to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to IMP administration;
* 17. Receipt of blood products within 2 months prior to SCR;
* 18. History of a major surgical procedure within 6 months prior to SCR. (NOTE: subjects may have had a cholecystectomy, provided not within 3 months of SCR and no complications with cholecystectomy);
* 19. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (eg, bariatric-metabolic surgery, etc.);
* 20. Poor peripheral venous access;
* 21. Known hypersensitivity to the IMP or any of its formulation excipients;
* 22. History or presence, upon clinical evaluation, of any illness that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results, or put the subject at undue risk;
* 23. Pregnancy or lactation;
* 24. Women of childbearing potential and non-sterile men who are not willing to use adequate contraception for the full duration of the study and for 90 days after the last dose of IMP.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-08-26 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration (Cmax) | Up to Day 9
  To evaluate pharmacokinetics (PK) following single and multiple ascending dose administration of G1090N in healthy subjects.
  Plasma PK parameters will be determined for tizoxanide (TZ) and tizoxanide glucuronide (TZG) concentrations including but not limited to Cmax.
Time to Cmax (tmax) | Up to Day 9
  To evaluate PK following single and multiple ascending dose administration of G1090N in healthy subjects.
  Plasma PK parameters will be determined for TZ and TZG concentrations including but not limited to tmax.
Area under the plasma concentration-time curve (AUC) | Up to Day 9
  To evaluate PK following single and multiple ascending dose administration of G1090N in healthy subjects.
  Plasma PK parameters will be determined for TZ and TZG concentrations including but not limited to AUC.
Terminal half-life (t1/2) | Up to Day 9
  To evaluate PK following single and multiple ascending dose administration of G1090N in healthy subjects.
  Plasma PK parameters will be determined for TZ and TZG concentrations including but not limited to t1/2.
Amount excreted (Ae) | Up to Day 8
  To evaluate PK following single and multiple ascending dose administration of G1090N in healthy subjects.
  Urine PK parameters will be determined for TZ and TZG concentrations including but not limited to Ae.
Renal clearance (CLr) | Up to Day 8
  To evaluate PK following single and multiple ascending dose administration of G1090N in healthy subjects.
  Urine PK parameters will be determined for TZ and TZG concentrations including but not limited to CLr.
Fraction of dose excreted (fe) | Up to Day 8
  To evaluate PK following single and multiple ascending dose administration of G1090N in healthy subjects.
  Urine PK parameters will be determined for TZ and TZG concentrations including but not limited to fe.

SECONDARY OUTCOMES:
To evaluate safety and tolerability following single and multiple ascending dose administration of G1090N in healthy subjects | from baseline up to Day 14
  Observed values and change from baseline, when relevant, for clinical laboratory safety parameters, vital signs measurements, 12-lead ECG parameters, and physical examinations.
  Safety and tolerability defined as the incidence and severity (NCI CTCAE v5.0 grade) of TEAEs including SAEs (comprising clinically significant findings on vital signs, physical examination, ECG, and laboratory parameters including change from baseline).

CONTACTS AND LOCATIONS:
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States